CLINICAL TRIAL: NCT05166499
Title: HMB Enriched Amino Acids to Reverse Muscle Loss in Cirrhosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Srinivasan Dasarathy, Staff, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-830
Record Dates: First submitted 2021-12-08; First posted 2021-12-22 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis | interventions — beta-hydroxyisovaleric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxy Methyl Butyrate (Active Comparator)
  Interventions: Dietary Supplement: Hydroxy Methyl Butyrate
- Balanced Amino Acid Mixture (Other)
  Interventions: Dietary Supplement: Balanced Amino Acids

INTERVENTIONS:
Dietary Supplement: Hydroxy Methyl Butyrate — Hydroxy Methyl Butyrate
  Arms: Hydroxy Methyl Butyrate
Dietary Supplement: Balanced Amino Acids — Balanced Amino Acids
  Arms: Balanced Amino Acid Mixture

SUMMARY:
Loss of skeletal muscle mass or sarcopenia is the most common and potentially reversible complication in cirrhosis that increases morbidity and mortality before, during and after liver transplantation. No proven treatments exist for the prevention or reversal of sarcopenia in cirrhosis, primarily because the mechanisms responsible for this are unknown. Based on compelling preliminary studies and those of the co investigator, investigators hypothesize that the mechanism of reduced skeletal muscle mass in cirrhosis is due to a myostatin mediated impaired mTOR (mechanistic target of rapamycin) signaling resulting in reduced protein synthesis and increased autophagy. Investigators further postulate that leucine, a direct stimulant of mTOR, will reverse the impaired mTOR phosphorylation in the skeletal muscle of cirrhotics. The consequent increase in protein synthesis reduced autophagy will result in an increase in skeletal muscle mass. Investigators will test these hypotheses by quantifying the response to acute and long term (3 month) administration of hydroxymethyl butyrate (HMB) enriched essential amino acid compared with an isonitrogenous isocaloric non-essential balanced amino acid mixture (does not stimulate protein synthesis) in cirrhotic patients. Fractional protein synthesis rate (FSR) in skeletal muscle, responses of the molecular regulatory pathways of skeletal muscle protein synthesis, and autophagy flux will be quantified in the acute and long term protocols. Tracer studies using L-[D5]-phenylalanine (Phe) as a primed constant infusion (prime 2µmol.kg-1.hr-1; constant 0.05 µmol.kg-1.hr-1) with and L [ring-D2] tyrosine, forearm plethysmography, and sequential skeletal muscle biopsies (total of 3 per study subject) will be used to quantify these outcomes. Anthropometric, clinical and body composition measures will be additional outcome measures for the long term intervention. Expression of regulatory signaling proteins, myostatin, IGF-1 (insulin like growth factor) , phospho-Akt, phospho-AMPK (activated protein kinase), phospho-mTOR and phospho-p70s6k will be quantified by Western immunoblots. Autophagy flux will be measured by quantifying expression of the autophagosome proteins.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cirrhosis of the liver
* Child-Pugh score of 5-8

Exclusion Criteria:

* Recent gastrointestinal bleeding (<3m)
* Active infection
* Overt encephalopathy
* Renal failure on dialysis
* Pedal edema
* Uncontrolled diabetes (HbA1C > 7.9mg/dL)
* Advanced cardiac, lung, kidney disease
* Metastatic cancer
* Medications that alter muscle protein metabolism
* Pregnancy
* Recent bowel resection or gastric bypass surgery,
* INR >1.7, platelets <60,000/ml, serum creatinine >2mg/dL
* Medications that interfere with blood clotting

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Fractional Synthesis Rate of Skeletal Muscle | Day 0 to Day 90
  To test whether fractional synthesis of skeletal muscle proteins changes from baseline to 90 days with the administration of BAA or EAA/LEU. Fractional synthesis rate (FSR) of mixed muscle proteins will be calculated from the incorporation rate of the L- [ring D5] phenylalanine into the proteins and the free tissue phenylalanine enrichments using precursor product model: FSR= (∆Ep/t)/(∆Ec) x60x100 and expressed as %/hour. ΔEp is the increment in myofibrillar protein-bound L- [ring D5] phenylalanine enrichment, t is the time between the muscle biopsies. ∆Ec is the L- [ring D5] phenylalanine enrichments in the free intracellular pool in the muscle biopsies.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States